CLINICAL TRIAL: NCT02506595
Title: A Pilot Randomized Controlled Trial of Treatment for Trauma-Related Nightmares Compared to Waitlist Control in Active Duty Military Personnel
Brief Title: A Trial of Treatment for Trauma-Related Nightmares in Active Duty Military Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 119-FP-15; HSC20150396H (Other: UTHSCSA IRB)
Record Dates: First submitted 2015-06-29; First posted 2015-07-23 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Nightmares

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ERRT-M for Nightmares (Experimental): Exposure, Relaxation, and Rescripting Therapy Military version (ERRT-M) -
  Interventions: Behavioral: ERRT-M for Nightmares
- Waitlist control (No Intervention): Participants randomized to the Waitlist control condition will be contacted once weekly for 5 weeks to monitored status and then invited to participant in treatment.

INTERVENTIONS:
Behavioral: ERRT-M for Nightmares — Exposure, Relaxation, and Rescripting Therapy Military version (ERRT-M) - Five 60-90 minute sessions administered once weekly. ERRT-M includes psychoeducation, sleep habit modification, relaxation training, written exposure to and rescription of nightmare content and imagery rehearsal of rescripted dream content.
  Other Names: Exposure Relaxation & Rescripting
  Arms: ERRT-M for Nightmares

SUMMARY:
The purpose of this study is to obtain preliminary data of the efficacy of Exposure, Relaxation, and Rescripting Therapy for nightmares among active duty military personnel.

DETAILED DESCRIPTION:
This will be a pilot randomized controlled trial to compare the effects of Exposure, Relaxation, and Rescripting Therapy for military populations (ERRT-M) among active duty service members. Participants will be randomized to 5 sessions of ERRT-M (n = 20 ) or to a 5-week waitlist control group (WL; n = 20).

Participants will complete all interviews and self-report measures 1 weeks following treatment or the WL condition and 1 month after completing treatment.

ELIGIBILITY:
Inclusion Criteria:

* Active duty military stationed at Fort Hood as assessed by self-report.
* Able to speak and read English.
* History of a traumatic event.
* Nightmare Disorder
* Stable on psychotropic and/or hypnotic medications and/or interventions for sleep (e.g., Continuous Positive Air Pressure for sleep apnea) administered by other providers for at least one month assessed by self-report and review of medical record.
* Willingness to refrain from beginning new behavioral health or medication treatment for issues pertaining to sleep, PTSD, or nightmares during participation in the study.
* Indication that the SM plans to be in the area for the 5 months following the first assessment

Exclusion Criteria:

* Current suicide or homicide risk meriting crisis intervention.
* Severe brain damage, assessed by the inability to comprehend baseline questionnaires.
* Pregnancy at baseline.
* Serious mental health diagnosis such as bipolar disorder or psychosis, assessed with the pre-treatment health interview and review of medical record.
* Currently taking propranolol.
* Currently engaged in evidence-based treatment for PTSD (i.e., Prolonged Exposure Therapy or Cognitive Processing Therapy) or Insomnia (i.e., Cognitive Behavioral Therapy for Insomnia).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of nightmares reported on the Nightmare Log | Change from baseline to 2-week posttreatment

SECONDARY OUTCOMES:
Total score on the Insomnia Severity Index (ISI) | Change from baseline to 2-week posttreatment
Total score on the Clinician Administered PTSD Scale (CAPS-5) | Change from baseline to 2-week posttreatment
Total score on the PTSD Checklist -DSM-5 (PCL-5) | Change from baseline to 2-week posttreatment
Total score on the Patient Health Questionnaire (PHQ-9) | Change from baseline to 2-week posttreatment

CONTACTS AND LOCATIONS:
Locations (1):
- Carl R Darnall Army Medical Center, Fort Hood, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pruiksma KE, Taylor DJ, Mintz J, Nicholson KL, Rodgers M, Young-McCaughan S, Hall-Clark BN, Fina BA, Dondanville KA, Cobos B, Wardle-Pinkston S, Litz BT, Roache JD, Peterson AL; STRONG STAR Consortium. A pilot randomized controlled trial of cognitive behavioral treatment for trauma-related nightmares in active duty military personnel. J Clin Sleep Med. 2020 Jan 15;16(1):29-40. doi: 10.5664/jcsm.8116. Epub 2019 Nov 26. PMID 31957648